CLINICAL TRIAL: NCT05706480
Title: Assessment of Gingival Thickness Using Colored Periodontal Probe Assessment Method: A Cross-Sectional Study
Brief Title: Assessment of Gingival Thickness Using Colored Periodontal Probe
Status: Completed | Type: Observational
Sponsor: Misr International University (Other)
Responsible Party: Sponsor
Other Study IDs: PER 4261006
Record Dates: First submitted 2023-01-23; First posted 2023-01-31 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-11

CONDITIONS: Gingival Phenotype
Keywords: Gingival thickness; Colored periodontal probe (CPP); Standard periodontal probe (SPP); Trans gingival sounding

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Periodontally clinically healthy patients: In Periodontally clinically healthy patients fulfilling the eligibility criteria. The gingival tissue thickness will be measured using probe-colored periodontal probes (CPP), standard periodontal probes (SPP) and transgingival sounding with an endodontic file (ISO #20), visual judgment using photographs will be done to the three assessment methods
  Interventions: Diagnostic Test: colored periodontal probes (CPP); Diagnostic Test: standard periodontal probes (SPP); Diagnostic Test: transgingival sounding with an endodontic file

INTERVENTIONS:
Diagnostic Test: colored periodontal probes (CPP) — The CPP will be placed with a force of approximately 0.2 N into the sulcus at the mid buccal surface of the tooth and the color that will be apparent from the tissue will be recorded
Diagnostic Test: standard periodontal probes (SPP) — The SPP (William's graduated probe) will be placed with a force of approximately 0.2 N into the sulcus at the mid buccal surface of the tooth and the color that will be apparent from the tissue will be recorded
Diagnostic Test: transgingival sounding with an endodontic file — the gingival thickness using the transgingival sounding. After application of local anesthesia gel an endodontic file (ISO 20) with a rubber stopper will be inserted perpendicularly into the buccal aspect of the gingiva (1 mm below the gingival margin) until it touches the tooth surface. The insertion depth will be ensured through placing the rubber stopper in contact with the gingiva and fixing its position and the distance between the tip and the rubber stopper will be calibrated using a manual calibration device (endodontic ruler).

SUMMARY:
the accuracy of different assessment methods of the gingival tissue thickness can be controversial affecting their correct classification and the techniques of gingival tissue management in case of mucogingival problems.

Aim: The aim of this study is to evaluate the accuracy of different assessment methods of measuring GT and to classify into the different gingival phenotypes.

DETAILED DESCRIPTION:
The accuracy of different assessment methods of the gingival tissue thickness can be controversial affecting their correct classification and the techniques of gingival tissue management in case of mucogingival problems.

The aim of this study is to evaluate the accuracy of different assessment methods of measuring GT and to classify into the different gingival phenotypes.

Periodontally clinically healthy patients will be recruited from the Dental Clinic Complex (MIU) according to eligibility criteria. The gingival tissue thickness will be measured using probe-colored periodontal probes (CPP), standard periodontal probes (SPP) and transgingival sounding with an endodontic file (ISO #20), visual judgment using photographs will be done to the three assessment methods. All readings including GT (1ry outcome) as well as keratinized tissue width and probing depth will be carried out by three calibrated outcome assessors. Data collected will be tabulated and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Systemically free patients (American Society of Anesthesiologists (ASA) I or II)
* Patients having a state of clinical periodontal health
* Patients aged from 18 to 65 years old
* Both genders
* Presence of anterior teeth in mandible and maxilla.
* Good oral hygiene

Exclusion Criteria:

* Carious teeth, teeth with crowns or veneers and non-carious cervical lesions
* Patients with healthy reduced periodontium.
* Smokers
* Pregnant and lactating females
* Patients taking drugs that affect the gingival tissues

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Periodontally clinically healthy patients, aged from 18 to 65 years old, with the presence of anterior teeth in mandible and maxilla and good oral hygiene
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
gingival thickness | baseline
  determination of the thickness of the gingival tissues

SECONDARY OUTCOMES:
Keratinized tissue width | baseline
  measuring the width of the keratinized tissue width in mm
Probing depth | baseline
  measuring of the distance from the gingival margin to the base of the pocket in mm

CONTACTS AND LOCATIONS:
Overall Officials: Zainab Hafez, Lecturer, Principal Investigator — Lecturer, faculty of oral and dental medicine misr international university; Shahinaz Al ashiry, Asso. Prof, Study Director — Associate professor, faculty of oral and dental medicine misr international university; Yahia Hassan, Lecturer, Principal Investigator — Lecturer, faculty of oral and dental medicine misr international universit
Locations (1):
- Faculty of oral and dental medicine, Misr international university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided